CLINICAL TRIAL: NCT02043080
Title: CIDRZ 1201 - Optimizing Clinical Outcomes in HIV-Infected Adults & Children Using Xpert MTB/RIF in Zambia
Brief Title: Optimizing Clinical Outcomes in HIV-Infected Adults & Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-1402
Record Dates: First submitted 2014-01-16; First posted 2014-01-23 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-05

CONDITIONS: Tuberculosis Diagnosis; HIV
Keywords: Tuberculosis; HIV; Xpert MTB/RIF; Determine TB-LAM; UNC; Zambia; Cost Effectiveness Analysis Curve; Centre for Infectious Disease Research in Zambia
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SOC: sputum smear and Chest x-ray (No Intervention): HIV-infected adult and pediatric TB suspects screened for TB according to current standard of care
- Xpert MTB/RIF, sputum, chest xray &TB culture (Experimental): HIV-infected adult and pediatric TB suspects screened for TB using the Xpert MTB/RIF Tuberculosis diagnostic tool (algorithm) which include chest x-ray, sputum TB culture
  Interventions: Other: Xpert MTB/RIF Tuberculosis diagnostic tool

INTERVENTIONS:
Other: Xpert MTB/RIF Tuberculosis diagnostic tool — This is s new diagnostic tool that has been approved by WHO for the diagnosis of TB in HIV-infected patients in resource limited settings
  Other Names: Gene Xpert MTB RIF (Cepheid Inc)
  Arms: Xpert MTB/RIF, sputum, chest xray &TB culture

SUMMARY:
This is a study to evaluate Xpert MTB/RIF as the first-line TB diagnostic test in HIV-infected adults and pediatric patients as a means to obtain faster, more accurate TB diagnosis.

DETAILED DESCRIPTION:
This study will evaluate Xpert Mycobacterium Tuberculosis/Rifampicin (MTB/RIF) as the first-line Tuberculosis (TB) diagnostic test in Human Immunodeficiency Virus (HIV)-infected adults and pediatric patients in peri-urban settings and determine its impact on accurate case detection and treatment initiation in these settings. In addition, the Determine TB-Lipoarabinomannan (LAM) Ag® will be used to model added diagnostic value when used alone or in combination with Xpert MTB/RIF, within the TB diagnostic algorithm for HIV infected patients in Zambia.

A quasi-experimental "before-after" study design will be used at two similar peri-urban district hospitals. Each site will initially implement the Standard of Care (SOC) phase, in which a prospective cohort of HIV-infected adult and pediatric TB suspects will be screened for TB according to the current standard of care in Zambian HIV care clinics. This will be followed by a 4-week "intervention wash-out" period to allow completion of the diagnostic work-up of all patients recruited during the last month of the SOC phase.

The second phase (Xpert MTB/RIF phase) will start immediately following the "intervention wash-out" period. In this phase, a second cohort of HIV-infected adult and pediatric TB suspects will be screened for TB using the Xpert MTB/RIF algorithm. Each phase will last approximately 6 months, or until the target sample size for adults is reached. Mycobacterial culture will be performed during the study to confirm TB diagnosis and determine whether appropriate treatment was given. "Appropriate treatment" means the patient was initiated on ATT within 4 weeks of screening initiation for culture-positive patients or a correct diagnosis of not having TB in culture-negative patients. Culture results will be released from the CIDRZ Lab for patient care as soon as results are available.

During both study phases participants will be asked to submit a urine sample for testing with the Determine TB-LAM Ag® assay. Urine specimens will be collected at the study site and all procedures will be carried out at the CIDRZ Central Laboratory in Lusaka using standard laboratory protocols and quality assurance procedures. Since Determine TB-LAM Ag® has not yet been endorsed by the World Health Organization (WHO) nor approved by the Zambian Ministry of Health for TB diagnosis, results from the Determine TB-LAM Ag® assay will not be used for patient care.

ELIGIBILITY:
Inclusion Criteria:

* Aged 15 years or above ("Adult"), or less than 15 years old ("Child") ;
* HIV-infected and enrolled in HIV care at Chongwe and Kafue District Hospitals
* Intends to continue receiving care at the district hospital for at least 6 months.
* TB suspects according to Zambian National Guidelines [31] ;
* Willing to provide signed informed consent (or parental consent, if the participant is under 18);
* Willing (or parent or guardian willing) to provide locator information and allow contact by phone or home visit

Exclusion Criteria:

* Diagnosed with TB within the last 6 months or taken TB treatment in the last 3 months
* Enrolled in another study which might interfere with study objectives (ex. TB-HAART)

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1436 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Proportions of adult and paediatric patients receiving appropriate TB treatment in each study phase | within 4 weeks of initiation
  proportions of adult and pediatric patients receiving appropriate TB treatment in each study phase, using mycobacterial culture as the reference standard, and the feasibility and cost effectiveness of Xpert MTB/RIF in this setting

SECONDARY OUTCOMES:
Clinical outcomes of subjects screened using the Xpert MTB/RIF algorithm compared to existing standard of care. | 3 and 6 months post TB-screening
  Clinical outcomes to be compared include (but are not limited to):
  ART treatment start date CD4 response TB treatment outcomes at 6 months post-diagnosis Mortality Co-morbidities Other Opportunistic Infections Characteristics of TB patients who initially test Xpert negative (Xpert- /Culture + patients)

OTHER OUTCOMES:
Diagnostic performance of Xpert MTB/RIF | screening visit, 3 and 6 months post screening
  Sensitivity, specificity, positive and negative predictive values of TB diagnosis with Xpert MTB/RIF compared to culture will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Stewart Reid, MD, Principal Investigator — University of North Carolina
Locations (1):
- Centre for Infectious Disease Research in Zambia, Lusaka, Zambia

REFERENCES:
- [Background] World Health Organization, Global Tuberculosis Control: WHO Report 2011. 2011:Geneva, Switzerland.
- [Background] Ayles H, Schaap A, Nota A, Sismanidis C, Tembwe R, De Haas P, Muyoyeta M, Beyers N; Peter Godfrey-Faussett for the ZAMSTAR Study Team. Prevalence of tuberculosis, HIV and respiratory symptoms in two Zambian communities: implications for tuberculosis control in the era of HIV. PLoS One. 2009;4(5):e5602. doi: 10.1371/journal.pone.0005602. Epub 2009 May 19. PMID 19440346
- [Background] Reid, S.E., Unpublished Data: Enhanced TB Screening to determine the prevalence and incidence of TB in a cohort of HIV clinic patients in Lusaka, Zambia. 2012.
- [Background] Lawn SD, Harries AD, Anglaret X, Myer L, Wood R. Early mortality among adults accessing antiretroviral treatment programmes in sub-Saharan Africa. AIDS. 2008 Oct 1;22(15):1897-908. doi: 10.1097/QAD.0b013e32830007cd. PMID 18784453
- [Background] Lawn SD, Kranzer K, Wood R. Antiretroviral therapy for control of the HIV-associated tuberculosis epidemic in resource-limited settings. Clin Chest Med. 2009 Dec;30(4):685-99, viii. doi: 10.1016/j.ccm.2009.08.010. PMID 19925961
- [Background] Henostroza, G., Unpublished work: Enhancing TB Screening in Zambian Prisons. 2011.
- [Background] Reid MJ, Shah NS. Approaches to tuberculosis screening and diagnosis in people with HIV in resource-limited settings. Lancet Infect Dis. 2009 Mar;9(3):173-84. doi: 10.1016/S1473-3099(09)70043-X. PMID 19246021
- [Background] Dawson R, Masuka P, Edwards DJ, Bateman ED, Bekker LG, Wood R, Lawn SD. Chest radiograph reading and recording system: evaluation for tuberculosis screening in patients with advanced HIV. Int J Tuberc Lung Dis. 2010 Jan;14(1):52-8. PMID 20003695
- [Background] Walls T, Shingadia D. Global epidemiology of paediatric tuberculosis. J Infect. 2004 Jan;48(1):13-22. doi: 10.1016/s0163-4453(03)00121-x. PMID 14667788
- [Background] Hesseling AC, Cotton MF, Jennings T, Whitelaw A, Johnson LF, Eley B, Roux P, Godfrey-Faussett P, Schaaf HS. High incidence of tuberculosis among HIV-infected infants: evidence from a South African population-based study highlights the need for improved tuberculosis control strategies. Clin Infect Dis. 2009 Jan 1;48(1):108-14. doi: 10.1086/595012. PMID 19049436
- [Background] Lawn SD. Point-of-care detection of lipoarabinomannan (LAM) in urine for diagnosis of HIV-associated tuberculosis: a state of the art review. BMC Infect Dis. 2012 Apr 26;12:103. doi: 10.1186/1471-2334-12-103. PMID 22536883
- [Background] Lusaka Urban District Health Management Team, Annual Tuberculosis Report. 2009.
- [Background] Turnbull ER, Kaunda K, Harris JB, Kapata N, Muvwimi MW, Kruuner A, Henostroza G, Reid SE. An evaluation of the performance and acceptability of three LED fluorescent microscopes in Zambia: lessons learnt for scale-up. PLoS One. 2011;6(11):e27125. doi: 10.1371/journal.pone.0027125. Epub 2011 Nov 4. PMID 22073271
- [Background] Kang'ombe CT, Harries AD, Ito K, Clark T, Nyirenda TE, Aldis W, Nunn PP, Semba RD, Salaniponi FM. Long-term outcome in patients registered with tuberculosis in Zomba, Malawi: mortality at 7 years according to initial HIV status and type of TB. Int J Tuberc Lung Dis. 2004 Jul;8(7):829-36. PMID 15260273
- [Background] Abdool Karim SS, Naidoo K, Grobler A, Padayatchi N, Baxter C, Gray A, Gengiah T, Nair G, Bamber S, Singh A, Khan M, Pienaar J, El-Sadr W, Friedland G, Abdool Karim Q. Timing of initiation of antiretroviral drugs during tuberculosis therapy. N Engl J Med. 2010 Feb 25;362(8):697-706. doi: 10.1056/NEJMoa0905848. PMID 20181971
- [Background] Blanc, F.-X., et al., Early (2 weeks) vs. late (8 weeks) initiation of highly active antiretroviral treatment (HAART) significantly enhance survival of severely immunosuppressed HIV-infected adults with newly diagnosed tuberculosis: results of the CAMELIA clinical trial. BMC Proceedings, 2011. 5(Suppl 1): p. O11.
- [Background] Havlir DV, Kendall MA, Ive P, Kumwenda J, Swindells S, Qasba SS, Luetkemeyer AF, Hogg E, Rooney JF, Wu X, Hosseinipour MC, Lalloo U, Veloso VG, Some FF, Kumarasamy N, Padayatchi N, Santos BR, Reid S, Hakim J, Mohapi L, Mugyenyi P, Sanchez J, Lama JR, Pape JW, Sanchez A, Asmelash A, Moko E, Sawe F, Andersen J, Sanne I; AIDS Clinical Trials Group Study A5221. Timing of antiretroviral therapy for HIV-1 infection and tuberculosis. N Engl J Med. 2011 Oct 20;365(16):1482-91. doi: 10.1056/NEJMoa1013607. PMID 22010914
- [Background] Nicol MP, Zar HJ. New specimens and laboratory diagnostics for childhood pulmonary TB: progress and prospects. Paediatr Respir Rev. 2011 Mar;12(1):16-21. doi: 10.1016/j.prrv.2010.09.008. Epub 2010 Oct 16. PMID 21172670
- [Background] Osborne CM. The challenge of diagnosing childhood tuberculosis in a developing country. Arch Dis Child. 1995 Apr;72(4):369-74. doi: 10.1136/adc.72.4.369. No abstract available. PMID 7763076
- [Background] Chintu C, Mudenda V, Lucas S, Nunn A, Lishimpi K, Maswahu D, Kasolo F, Mwaba P, Bhat G, Terunuma H, Zumla A; UNZA-UCLMS Project Paediatric Post-mortem Study Group. Lung diseases at necropsy in African children dying from respiratory illnesses: a descriptive necropsy study. Lancet. 2002 Sep 28;360(9338):985-90. doi: 10.1016/S0140-6736(02)11082-8. PMID 12383668
- [Background] World Health Organization, Roadmap for rolling out Xpert MTB/RIF for rapid diagnosis of TB and MDR-TB. 2010.
- [Background] Boehme CC, Nabeta P, Hillemann D, Nicol MP, Shenai S, Krapp F, Allen J, Tahirli R, Blakemore R, Rustomjee R, Milovic A, Jones M, O'Brien SM, Persing DH, Ruesch-Gerdes S, Gotuzzo E, Rodrigues C, Alland D, Perkins MD. Rapid molecular detection of tuberculosis and rifampin resistance. N Engl J Med. 2010 Sep 9;363(11):1005-15. doi: 10.1056/NEJMoa0907847. Epub 2010 Sep 1. PMID 20825313
- [Background] Hillemann D, Rusch-Gerdes S, Boehme C, Richter E. Rapid molecular detection of extrapulmonary tuberculosis by the automated GeneXpert MTB/RIF system. J Clin Microbiol. 2011 Apr;49(4):1202-5. doi: 10.1128/JCM.02268-10. Epub 2011 Jan 26. PMID 21270230
- [Background] Nicol MP, Workman L, Isaacs W, Munro J, Black F, Eley B, Boehme CC, Zemanay W, Zar HJ. Accuracy of the Xpert MTB/RIF test for the diagnosis of pulmonary tuberculosis in children admitted to hospital in Cape Town, South Africa: a descriptive study. Lancet Infect Dis. 2011 Nov;11(11):819-24. doi: 10.1016/S1473-3099(11)70167-0. Epub 2011 Jul 19. PMID 21764384
- [Background] Policy Statement: Automated Real-Time Nucleic Acid Amplification Technology for Rapid and Simultaneous Detection of Tuberculosis and Rifampicin Resistance: Xpert MTB/RIF System. Geneva: World Health Organization; 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK304235/ PMID 26158191
- [Background] Boehme CC, Nicol MP, Nabeta P, Michael JS, Gotuzzo E, Tahirli R, Gler MT, Blakemore R, Worodria W, Gray C, Huang L, Caceres T, Mehdiyev R, Raymond L, Whitelaw A, Sagadevan K, Alexander H, Albert H, Cobelens F, Cox H, Alland D, Perkins MD. Feasibility, diagnostic accuracy, and effectiveness of decentralised use of the Xpert MTB/RIF test for diagnosis of tuberculosis and multidrug resistance: a multicentre implementation study. Lancet. 2011 Apr 30;377(9776):1495-505. doi: 10.1016/S0140-6736(11)60438-8. Epub 2011 Apr 18. PMID 21507477
- [Background] Marlowe EM, Novak-Weekley SM, Cumpio J, Sharp SE, Momeny MA, Babst A, Carlson JS, Kawamura M, Pandori M. Evaluation of the Cepheid Xpert MTB/RIF assay for direct detection of Mycobacterium tuberculosis complex in respiratory specimens. J Clin Microbiol. 2011 Apr;49(4):1621-3. doi: 10.1128/JCM.02214-10. Epub 2011 Feb 2. PMID 21289151
- [Background] Theron G, Peter J, van Zyl-Smit R, Mishra H, Streicher E, Murray S, Dawson R, Whitelaw A, Hoelscher M, Sharma S, Pai M, Warren R, Dheda K. Evaluation of the Xpert MTB/RIF assay for the diagnosis of pulmonary tuberculosis in a high HIV prevalence setting. Am J Respir Crit Care Med. 2011 Jul 1;184(1):132-40. doi: 10.1164/rccm.201101-0056OC. Epub 2011 Apr 14. PMID 21493734
- [Background] Lawn SD, Little F, Bekker LG, Kaplan R, Campbel E, Orrell C, Wood R. Changing mortality risk associated with CD4 cell response to antiretroviral therapy in South Africa. AIDS. 2009 Jan 28;23(3):335-42. doi: 10.1097/QAD.0b013e328321823f. PMID 19114870
- [Background] Badri M, Wilson D, Wood R. Effect of highly active antiretroviral therapy on incidence of tuberculosis in South Africa: a cohort study. Lancet. 2002 Jun 15;359(9323):2059-64. doi: 10.1016/S0140-6736(02)08904-3. PMID 12086758
- [Background] Zambia Ministry of Health National Tuberculosis and Leprosy Control Programme, Tuberculosis and TB/HIV Manual. 2008: Lusaka.
- [Background] World Health Organization, Rapid Implementation of the Xpert MTB/RIF diagnostic test: Technical and operational 'How-to' Practical considerations. 2011.
- [Background] Francis J. Curry National Tuberculosis Center Institutional Consultation Services, Conducting Sputum Induction Safely. 1999.
- [Background] World Health Organization, Guidelines for cost and cost-effectivness analysis of tuberculosis control. 2002.
- [Background] Petitti, D., Meta-Analysis, Decision Analysis, and Cost-Effectivness Analysis. Methods for Quantitative Synthesis in Medicine. 2nd edition ed. 2000, New York: Oxford Press.
- [Background] Drummond MF, S., M.J., Torrance, G.W., O'Brien, B.J., Stoddart, G.L., Methods for the Economic Evaluation of Health Car Programmes. Vol. 3rd edition. 2005: Oxford University Press.
- [Background] Craig BA, Black MA. Incremental cost-effectiveness ratio and incremental net-health benefit: two sides of the same coin. Expert Rev Pharmacoecon Outcomes Res. 2001 Oct;1(1):37-46. doi: 10.1586/14737167.1.1.37. PMID 19807506
- [Background] Hoch JS, Rockx MA, Krahn AD. Using the net benefit regression framework to construct cost-effectiveness acceptability curves: an example using data from a trial of external loop recorders versus Holter monitoring for ambulatory monitoring of "community acquired" syncope. BMC Health Serv Res. 2006 Jun 6;6:68. doi: 10.1186/1472-6963-6-68. PMID 16756680
- See also: University of North Carolina website — http://www.unc.edu